CLINICAL TRIAL: NCT06891885
Title: A Prospective, Open-label, Single-arm, Dose-escalation Study of the Safety and Tolerability of a Single Subretinal Uniocular Injection of Allogeneic Induced Pluripotent Stem Cell (iPSC)-Derived Retinal Sheets (DSP-3077) in Adults With Retinitis Pigmentosa (RP)
Brief Title: A Study to Investigate the Safety of DSP-3077 After a Unilateral Eye Injection in Male and Female Participants 18 Years of Age or Older With Retinitis Pigmentosa
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DE101101
Record Dates: First submitted 2025-02-27; First posted 2025-03-24 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa | interventions — KPNA1 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Experimental): Best Corrected Visual Acuity (BCVA) in the study eye between hand motion and 20 Early Treatment Diabetic Retinopathy Study (ETDRS) letter score (approximately ≤ 20/400 Snellen equivalent), inclusive at Screening and Baseline
  Interventions: Drug: DSP-3077 Retinal Sheet Cohort 1
- Cohort 2 (Experimental): Best Corrected Visual Acuity (BCVA) in the study eye between hand motion and 20 Early Treatment Diabetic Retinopathy Study (ETDRS) letter score (approximately ≤ 20/400 Snellen equivalent), inclusive at Screening and Baseline
  Interventions: Drug: DSP-3077 Retinal Sheet Cohort 2
- Cohort 3 (Experimental): Best Corrected Visual Acuity (BCVA) in the study eye between 20 Early Treatment Diabetic Retinopathy Study (ETDRS) letter score (approximately ≥ 20/400 Snellen equivalent) and 35 ETDRS letter score (approximately ≤ 20/200 Snellen equivalent), inclusive at Screening; BCVA in the study eye between 10 ETDRS letter score (approximately ≥ 20/640 Snellen equivalent) and 35 ETDRS letter score (approximately ≤ 20/200 Snellen equivalent) at Baseline
  Interventions: Drug: DSP-3077 Retinal Sheet Cohort 3

INTERVENTIONS:
Drug: DSP-3077 Retinal Sheet Cohort 1 — For each participant only 1 eye will receive a low dose (>= 0.8 to < 2.4 mm2) of single subretinal injection of DSP-3077 using the DSP-3077-delivery device on Day 1
  Other Names: Cohort 1
  Arms: Cohort 1
Drug: DSP-3077 Retinal Sheet Cohort 2 — For each participant only 1 eye will receive a high dose (>= 2.4 to < 6.4 mm2) of single subretinal injection of DSP-3077 using the DSP-3077-delivery device on Day 1
  Other Names: Cohort 2
  Arms: Cohort 2
Drug: DSP-3077 Retinal Sheet Cohort 3 — For each participant only 1 eye will receive a high dose (>= 2.4 to < 6.4 mm2) of single subretinal injection of DSP-3077 using the DSP-3077-delivery device on Day 1
  Other Names: Cohort 3
  Arms: Cohort 3

SUMMARY:
The Goal of this study is to evaluate the safety, tolerability, and clinical responses following single dose of DSP-3077. Study enrolls both male and female patients in 3 cohorts with each cohort defined by visual acuity (VA) criteria and dose level of DSP-3077. Each cohort will include 4 participants.

DETAILED DESCRIPTION:
This is a Phase 1/2a, open-label, single-arm, uncontrolled, dose-escalation study evaluating 2 dose levels of iPSC-derived retinal sheets (DSP-3077) administered with a single subretinal uniocular injection in adults with RP. The total duration of participant participation will be approximately 65 months from start of Screening through end of Extension Observation Period Part B. After an initial 2-week period of frequent visits after surgery, the visit frequency will be approximately monthly through Month 4, every 3 months through Month 24, and every 6 months through Month 60. After completion of Study DE101101 (Month 60 Visit or ET Visit) and under a separate process, the Sponsor will collect long-term data following treatment with DSP-3077, annually from 6 years to 15 years after DSP-3077 administration to further characterize the long-term safety of DSP-3077.

Participants will be treated in 3 cohorts, with each cohort defined by visual acuity (VA) criteria and dose level of DSP-3077. Each cohort will include 4 participants for a total of 12 participants.

Primary objective is to evaluate the safety and tolerability of 2 dose levels of DSP-3077 in adults with RP. Other objectives are to evaluate the safety, engraftment, and potential therapeutic response of 2 dose levels of DSP-3077 in adults with RP and to evaluate DSP-3077-delivery device performance.

ELIGIBILITY:
Inclusion Criteria:

* Participant is >= 18 years of age at the time of signing the informed consent.
* Participant has a clinical diagnosis of nonsyndromic retinitis pigmentosa.
* Participant is willing to consent to genetic testing, if not already done.
* Cohorts 1 and 2: Participant will have BCVA in the study eye between hand motion and 20 ETDRS letter score (approximately <= 20/400 Snellen equivalent), inclusive at Screening and Baseline.
* Cohort 3: Participant will have BCVA in the study eye between 20 ETDRS letter score (approximately >= 20/400 Snellen equivalent) and 35 ETDRS letter score (approximately <= 20/200 Snellen equivalent), inclusive at Screening.
* Participant is in good physical health, based on medical history, physical examination, vital signs, electrocardiogram (ECG), and clinical laboratory tests at Screening.

Exclusion Criteria:

* Participant has an eye disease or visual disorder other than RP that impairs visual function (eg, retinal vascular disease, glaucoma).
* Participant has any other eye condition (eg, ocular media opacity, nystagmus), which in the opinion of the investigator, would preclude an accurate evaluation at any time during the study and/or make surgical delivery more challenging.
* Participant has any clinically significant unstable medical condition or any clinically significant chronic disease that in the opinion of the investigator, would limit the participant's ability to complete and/or participate in the study.
* Female participant who is pregnant or lactating or planning to become pregnant.
* Participant has received treatment with any nonapproved, experimental, or investigational therapy in either eye (systemic, topical, intravitreal) and/or received treatment in an interventional clinical trial for an eye disease or disorder within 90 days or 5 half-lives, whichever is longer, prior to Screening.
* Participant has previously received cell therapy, gene augmentation therapy, genome editing therapy, or any subretinal administered therapy for an eye disease or disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-10-23 (Estimated); Primary Completion 2028-10-31 (Estimated); Study Completion 2032-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of ocular adverse events (AEs) | 60 months
Incidence of ocular serious adverse events (SAEs) | 60 months
Incidence of ocular adverse events (AEs) leading to discontinuation | 60 months
Incidence of adverse events (AEs) | 60 months
Incidence of serious adverse events (SAEs) | 60 months
Incidence of adverse events (AEs) leading to discontinuation | 60 months
Incidence of adverse events (AEs) leading to death | 60 months

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts Eye and Ear, Boston, Massachusetts, United States